CLINICAL TRIAL: NCT01474252
Title: Comparison of Intubation Duration Between Rapid Sequence Intubation Technique and Non- Rapid Sequence Intubation Technique in Siriraj Hospital by Emergency Medicine Residences
Brief Title: Comparison of Intubation Duration Between Rapid Sequence Intubation (RSI) Technique and Non-RSI Technique
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Mingkwan Wongyingsinn, MD, Assistant Professor, Siriraj Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: SIRB213
Record Dates: First submitted 2011-11-09; First posted 2011-11-18 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-06

CONDITIONS: Tracheal Intubation Morbidity
MeSH Terms: interventions — Rapid Sequence Induction and Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RSI technique (Experimental): Intubation with RSI technique. RSI technique includes the administration of inductive and neuromuscular blocking agents to facilitate an intubation.
  In this study, we have no restriction of medication use. Physicians can chose any of medication as an individual judgement.
  Interventions: Drug: RSI
- Non-RSI (No Intervention): Intubation without RSI technique. No any medication use during intubation period.

INTERVENTIONS:
Drug: RSI — All medications are administered only one dose before intubation
  Anesthetics:
  Propofol 2-2.5 mg/kg Thiopental 3-5mg/kg Etomidate 1-2mg/kg
  Neuromuscular blocking agents:
  Succinylcholine 1-1.5mg/kg Rocuronium 0.9mg/kg
  Opioid:
  Fentanyl 1-2ug/kg
  Other Names: Rapid Sequence Intubation
  Arms: RSI technique

SUMMARY:
The purpose of this study is to evaluate intubation duration between rapid sequence intubation technique (RSI) and non-rapid sequence intubation technique (non-RSI) performed by emergency medicine residents in Siriraj hospital.

DETAILED DESCRIPTION:
A prospective cohort study was conducted in the non-traumatic emergency department (ED).

ELIGIBILITY:
Inclusion Criteria:

* patients required airway control by tracheal intubation

Exclusion Criteria:

* cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2008-07; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The overall intubation duration | Participants will be followed for the overall intubation duration until confirmation the endotracheal position, an expected average of 2 minutes
  The overall intubation duration is recorded on the decision to intubation patient and corresponds to the time of confirmation the endotracheal position by chest auscultation

SECONDARY OUTCOMES:
the intubation duration | Participants will be followed for the intubation duration until confirmation the endotracheal position, an expected average of 5 minutes
  The intubation duration (Ti), it is defined from application the laryngoscope into the patient's mouth to the time of confirmation an endotracheal position
Complication | Participants will be followed in the period of staying in the emergency room and hospital, an expected average of 4 weeks
  Complications occur during and after intubation peroid are recorded and monitored until patients are discharged fromt the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Mingkwan Wongyingsinn, M.D., Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkok, Bangkok, Thailand